CLINICAL TRIAL: NCT03594786
Title: To Assess Hemodynamic Disturbances to the Ostia of the Renal Arteries Generated by the Implantation of EVAR With a Suprarenal Fixation
Brief Title: Impact of Supra-renal Fixation of EVAR on Hemodynamics of Renal Arteries
Acronym: IFIXEAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A03047-46
Record Dates: First submitted 2018-04-24; First posted 2018-07-20 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Aortic Aneurysm, Abdominal; Endovascular Procedures; Renal Artery Stenosis
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Renal Artery Obstruction | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- endovascular aneurysm repair (EVAR) arm (Experimental): every patients are in the same arm and have EVAR with supra-renal fixation
  Interventions: Device: endovascular aneurysm repair (EVAR)

INTERVENTIONS:
Device: endovascular aneurysm repair (EVAR) — Patient will be enrolled when the decision of an endovascular procedure with supra renal fixation is required. Before the intervention, Duplex scan will be necessary to evaluate renal arteries ostia. This exam will be realised in the month after the intervention and one year later.

SUMMARY:
The investigators conducted a bicentric prospective study to quantify the hemodynamic disturbances to the ostia of the renal arteries generated by the implantation EVAR with suprarenal fixation immediately postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* elective EVAR with supra renal fixation
* women who have been postmenopausal for at least 24 months or are surgically sterilized, or for women of childbearing potential, use of an effective method of contraception
* consent to participate
* Affiliation to a French social security

Exclusion Criteria:

* stenosis of at least one renal artery
* dialysis
* rupture of abdominal aortic aneurysm
* renal stenting during the procedure
* fenestrated EVAR
* legal incapacity or limited legal capacity
* subject being in the exclusion period of another study
* pregnant woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
systolic maximum speed at the ostia of the renal arteries | one month
  Quantify the hemodynamic disturbances to the ostia of the renal arteries generated by the implantation of a suprarenal fixation aortic stent immediately postoperatively.

SECONDARY OUTCOMES:
systolic maximum speed at the ostia of the renal arteries | one year
  Quantify the hemodynamic disturbances to the ostia of the renal arteries generated by the implantation of a suprarenal fixation aortic stent immediately postoperatively.
proportion of patients with renal artery stenosis | one year
proportion of disappearance of the "notch" (pre-systolic notch) | one year
proportion of increase in systolic rise time | one year
proportion of decrease of the resistance index | one year
proportion of post-stenotic turbulence | one year
glomerular filtration rate | one year
  estimation of the glomerular filtration rate calculated by CKD-EPI between the preoperative and at one year

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hosptalier Universitaire, Besançon
  - Centre Hospitalier Universitaire, Dijon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salomon du Mont L, Parmentier AL, Puyraveau M, Mauny F, Guillon B, Rinckenbach S, Costa P. To assess hemodynamic disturbances to the ostia of the renal arteries generated by the implantation of EVAR with a suprarenal fixation. Medicine (Baltimore). 2020 May;99(18):e19917. doi: 10.1097/MD.0000000000019917. PMID 32358359